CLINICAL TRIAL: NCT05315830
Title: A Single-Arm, Open-Label, Exploratory Study to Evaluate the Safety of HER2 Tumor Vaccine Injection Alone/in Combination With Standard of Care Chemotherapy in Patients With her2/Neu Overexpressing Metastatic or Advanced Adenocarcinoma of the Stomach or Gastroesophageal Junction
Brief Title: A Study of HER2 Tumor Vaccine in Patients With Her-2 Positive Gastric/GEJ Adenocarcinoma Esophagogastric
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Wang Zishu, MD，Head of Oncology Department, Principal Investigator, The First Affiliated Hospital of Bengbu Medical University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LWY22003CBY
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Adenocarcinoma - GEJ; Adenocarcinoma of the Stomach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HER2 Vaccine alone (Experimental): 0.6 μg HER2 Vaccine
  Interventions: Biological: HER2 Tumor Vaccine
- HER2 Vaccine plus Standard of Care Chemotherapy (Experimental): 0.6 μg HER2 Vaccine plus Cisplatin and either Fluorouracil (5-FU) or Capecitabine or other Standard of Care Chemotherapy
  Interventions: Biological: HER2 Tumor Vaccine+ Standard of Care chemotherapy

INTERVENTIONS:
Biological: HER2 Tumor Vaccine — B-cell epitope vaccine HER2 Tumor Vaccine 0.6 μg，Intramuscular injection on D1, D14 and D28
  Arms: HER2 Vaccine alone
Biological: HER2 Tumor Vaccine+ Standard of Care chemotherapy — B-cell epitope vaccine HER2 Tumor Vaccine 0.6 μg，Intramuscular injection on D1, D14 and D28 Standard of Care Chemotherapy cisplatin by intravenous administration at 80 mg/m2 on the first day of each cycle and either 5-FU, 4000 mg/m2 CIV (administered as 1000 mg/m2/day as continuous infusion for 96 hours on days 1 to 4 of each cycle) or capecitabine for 14 days at 2000 mg/m2/day, orally (administered as 1000 mg/m2 twice daily morning and evening for a total of 2000 mg/m2/day on days 1 to 14 of each cycle) or other standard of care chemotherapy
  Arms: HER2 Vaccine plus Standard of Care Chemotherapy

SUMMARY:
This is a single-arm, open-label, clinical study to evaluate the safety of HER2 tumor vaccine injection alone/in combination with standard of care chemotherapy in patients with HER2/neu overexpressing gastric or gastroesophageal junction (GEJ) adenocarcinoma.

The purpose of this study is to evaluate the safety and tolerability, antitumor activity, The immunoreactivity, pharmacokinetics and of HER2 tumor vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years;
* Metastatic gastric or GEJ adenocarcinoma, or locally advanced disease not amenable to surgical resection;
* HER2/neu overexpression (3+ by immunohistochemistry (IHC) or if IHC 2+ confirmed by fluorescent in situ hybridization [FISH];
* ECOG score of 0 ~ 2;
* Adequate bone marrow, hepatic and renal and coagulation function;
* Women of childbearing age who have a negative pregnancy test within 7 days before treatment. Female patients of childbearing age, and male patients with partners of childbearing age must agree to use at least one medically recognized contraceptive method during study treatment and within at least 6 months after the last dose of investigational drug;
* Voluntarily participated in this study, signed the informed；

Exclusion Criteria:

* Continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 4 weeks prior to first dose of study treatment. Inhaled or topical steroids and physiological replacement doses of up to 10 mg daily prednisone equivalents are permitted in the absence of active auto-immune disease；
* Subjects who have had major surgery within 4 weeks before HER2 tumor vaccine administration
* Subjects who have received anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, etc within 5 elimination half-life prior first dose of HER2 tumor vaccine treatment;
* Subjects with known brain metastasis and/or clinically history tumor brain of metastasis；
* Patients with uncontrollable pleural effusion, abdominal effusion and pericardial effusion;
* Active infection requiring treatment. HIV, HCV, syphilis, CMV, EBV infected patients; Patients with active HBV replication
* Other conditions that the investigator assessed as ineligible for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Graded according to the NCI CTCAE version 5.0.

SECONDARY OUTCOMES:
To evaluate the antitumor activity | Up to 2 years
  To assess per RECIST and iRECIST
Humoral and cellular immunogenicity of HER2 Tumor Vaccine | Up to 6 months
  Values and changes from randomization in humoral and cellular immunogenicity data including P467-specific antibodies (IgG), Her-2-specific antibodies (IgG), vaccine-specific cytokine levels and regulatory and effector T and B cells.

CONTACTS AND LOCATIONS:
Overall Officials: Zishu Wang, MD, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- First Affiliated Hospital Bengbu Medical College, Bengbu, Anhui, China